CLINICAL TRIAL: NCT05844098
Title: Arthroscopic Assisted CC Stabilization Alone VS Additional K-wire Fixation for Acute Acromioclavicular Joint Injury, A Randomized Controlled Trial
Brief Title: Arthroscopic Assisted CC Stabilization Alone VS Additional K-wire Fixation for Acute Acromioclavicular Joint Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Savang Vadhana Memorial Hospital, Thailand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Interventional
Record Dates: First submitted 2023-02-16; First posted 2023-05-06 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Acromioclavicular Joint Dislocation
Keywords: Arthroscopic assisted CC-stabilization; AC joint injury
MeSH Terms: interventions — Bone Wires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With K-wire (Experimental): arthroscopic assisted CC-stabilization with K-wire
  Interventions: Device: K-wire
- No K-wire (No Intervention): arthroscopic assisted CC-stabilization

INTERVENTIONS:
Device: K-wire — K-wire No. 2.0 insertion was done additionally from arthroscopic assisted CC-stabilization by inserting K-wire from acromion process to distal clavicle.
  Arms: With K-wire

SUMMARY:
This RCT study is designed for comparing functional outcomes and radioligic outcomes between intervention group (Arthroscopic assisted CC-stabilzation with additional K-wire fixation) and control group (Arthroscopic assisted CC-stabilzation alone) for acute ACJI.

The main question it aims to answer is:

- Does Arthroscopic assisted CC-stabilization with additional K-wire fixation provide different outcomes in functional outcomes, CC-distance and GACA difference compare with arthroscopic assisted CC-stabilization alone in acute acromioclavicular joint injury?

DETAILED DESCRIPTION:
Acromioclavicular joint injury (ACJI) is one of the most common injury of shoulder joint. Most common mechanism of injury is from direct force apply to the affected shoulder, in adduction position, in acromion process area. Most of the intervention that have been used for treat ACJI are focused on pain control, maintain the strength of the joint, no limitation in daily life activity and full range of motion of affected shoulder. Operative treatment is indicated in ACJI Rockwood classification grade III, IV, V, and VI. Nowadays there are over 60 surgical techniques without gold standard. Arthroscopic assisted CC-stabilzation is one of the most popular technique that has been used for ACJI.

This RCT study is designed for comparing functional outcomes (ACJI score, VAS, Constant score and DASH score) and radioligic outcomes (CC-distance difference, GACA difference) between intervention group (Arthroscopic assisted CC-stabilzation with additional K-wire fixation) and control group (Arthroscopic assisted CC-stabilzation alone) for acute ACJI.

The main question it aims to answer is:

- Does Arthroscopic assisted CC-stabilization with additional K-wire fixation provide different outcomes in functional outcomes, CC-distance and GACA difference compare with arthroscopic assisted CC-stabilization alone in acute acromioclavicular joint injury?

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45 years old
* Acute AC joint injury rockwood classification III, IV and V

Exclusion Criteria:

* History of underwent previous ipsilateral shoulder surgery
* Specific active associated ipsilateral injury (Rib fractures, clavicel fractures, scapula fractures and base of coracoid fractures)
* Onset of injury more than 3 weeks
* Cannot underwent arthroscopic assisted CC-stabilization surgery

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Acromioclavicular Joint Instability (ACJI) score | 1 year post-operative
  Functional outcome, Rated from 0-100, higher score means better function of the shoulder

SECONDARY OUTCOMES:
Coracoclavicular (CC) distance diference | Postoperative day 1, 2weeks postop, 6weeks postop, 3months postop, 6 months postop, 1 year postop
  Radiologic outcome
Gleno-acromio-clavicular angle (GACA) difference | 3months postop, 6 months postop, 1 year postop
  Radiologic outcome
Constant score | 3months postop, 6 months postop, 1 year postop
  Functional outcome, Score from 0-100, Higher score means better shoulder function
DASH score | 3months postop, 6 months postop, 1 year postop
  Functional outcome, Score from 0-100, 0 means no disabillity, 100 means most severe disabillity
VAS | 3months postop, 6 months postop, 1 year postop
  Functional outcome, Scale from 0-10, Lower score means better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Nachapong Sithiwichankit, MD, Principal Investigator — QSMVH
Locations (1):
- Queen Savang Vadhana Memorial Hospital, Chon Buri, Thailand

REFERENCES:
- [Background] Frank RM, Cotter EJ, Leroux TS, Romeo AA. Acromioclavicular Joint Injuries: Evidence-based Treatment. J Am Acad Orthop Surg. 2019 Sep 1;27(17):e775-e788. doi: 10.5435/JAAOS-D-17-00105. PMID 31008872
- [Background] Goldenberg MM. Analysis of the inhibitory innervation of the isolated gerbil colon. Arch Int Pharmacodyn Ther. 1968 Oct;175(2):347-64. No abstract available. PMID 5702953
- [Background] Beitzel K, Mazzocca AD, Bak K, Itoi E, Kibler WB, Mirzayan R, Imhoff AB, Calvo E, Arce G, Shea K; Upper Extremity Committee of ISAKOS. ISAKOS upper extremity committee consensus statement on the need for diversification of the Rockwood classification for acromioclavicular joint injuries. Arthroscopy. 2014 Feb;30(2):271-8. doi: 10.1016/j.arthro.2013.11.005. PMID 24485119
- [Background] Nolte PC, Lacheta L, Dekker TJ, Elrick BP, Millett PJ. Optimal Management of Acromioclavicular Dislocation: Current Perspectives. Orthop Res Rev. 2020 Mar 5;12:27-44. doi: 10.2147/ORR.S218991. eCollection 2020. PMID 32184680
- [Background] Aliberti GM, Kraeutler MJ, Trojan JD, Mulcahey MK. Horizontal Instability of the Acromioclavicular Joint: A Systematic Review. Am J Sports Med. 2020 Feb;48(2):504-510. doi: 10.1177/0363546519831013. Epub 2019 Apr 23. PMID 31013137
- [Background] Cisneros LN, Reiriz JS. Prevalence of remaining horizontal instability in high-grade acromioclavicular joint injuries surgically managed. Eur J Orthop Surg Traumatol. 2017 Apr;27(3):323-333. doi: 10.1007/s00590-016-1898-0. Epub 2017 Jan 5. PMID 28054147
- [Background] Shin SJ, Kim NK. Complications after arthroscopic coracoclavicular reconstruction using a single adjustable-loop-length suspensory fixation device in acute acromioclavicular joint dislocation. Arthroscopy. 2015 May;31(5):816-24. doi: 10.1016/j.arthro.2014.11.013. Epub 2014 Dec 25. PMID 25543250
- [Background] Tauber M, Koller H, Hitzl W, Resch H. Dynamic radiologic evaluation of horizontal instability in acute acromioclavicular joint dislocations. Am J Sports Med. 2010 Jun;38(6):1188-95. doi: 10.1177/0363546510361951. Epub 2010 Apr 1. PMID 20360606
- [Background] Minkus M, Hann C, Scheibel M, Kraus N. Quantification of dynamic posterior translation in modified bilateral Alexander views and correlation with clinical and radiological parameters in patients with acute acromioclavicular joint instability. Arch Orthop Trauma Surg. 2017 Jun;137(6):845-852. doi: 10.1007/s00402-017-2691-1. Epub 2017 Apr 17. PMID 28417201
- [Background] Cano-Martinez JA, Nicolas-Serrano G, Bento-Gerard J, Picazo-Marin F, Andres-Grau J. Acute high-grade acromioclavicular dislocations treated with triple button device (MINAR): Preliminary results. Injury. 2016 Nov;47(11):2512-2519. doi: 10.1016/j.injury.2016.09.029. Epub 2016 Sep 15. PMID 27663286
- [Background] Scheibel M, Droschel S, Gerhardt C, Kraus N. Arthroscopically assisted stabilization of acute high-grade acromioclavicular joint separations. Am J Sports Med. 2011 Jul;39(7):1507-16. doi: 10.1177/0363546511399379. Epub 2011 Mar 24. PMID 21436458
- [Background] Sumanont S, Nopamassiri S, Boonrod A, Apiwatanakul P, Boonrod A, Phornphutkul C. Acromioclavicular joint dislocation: a Dog Bone button fixation alone versus Dog Bone button fixation augmented with acromioclavicular repair-a finite element analysis study. Eur J Orthop Surg Traumatol. 2018 Aug;28(6):1095-1101. doi: 10.1007/s00590-018-2186-y. Epub 2018 Mar 20. PMID 29557509
- [Background] Ladermann A, Grosclaude M, Lubbeke A, Christofilopoulos P, Stern R, Rod T, Hoffmeyer P. Acromioclavicular and coracoclavicular cerclage reconstruction for acute acromioclavicular joint dislocations. J Shoulder Elbow Surg. 2011 Apr;20(3):401-8. doi: 10.1016/j.jse.2010.08.007. PMID 20888260
- [Background] Cho CH, Kim BS, Kwon DH. Importance of additional temporary pin fixation combined coracoclavicular augmentation using a suture button device for acute acromioclavicular joint dislocation. Arch Orthop Trauma Surg. 2016 Jun;136(6):763-70. doi: 10.1007/s00402-016-2437-5. Epub 2016 Mar 10. PMID 26965695
- [Background] Vrgoc G, Japjec M, Jurina P, Gulan G, Jankovic S, Sebecic B, Staresinic M. Operative treatment of acute acromioclavicular dislocations Rockwood III and V-Comparative study between K-wires combined with FiberTape((R)) vs. TightRope System((R)). Injury. 2015 Nov;46 Suppl 6:S107-12. doi: 10.1016/j.injury.2015.10.053. Epub 2015 Nov 14. PMID 26584732
- [Background] Dyrna F, Imhoff FB, Haller B, Braun S, Obopilwe E, Apostolakos JM, Morikawa D, Imhoff AB, Mazzocca AD, Beitzel K. Primary Stability of an Acromioclavicular Joint Repair Is Affected by the Type of Additional Reconstruction of the Acromioclavicular Capsule. Am J Sports Med. 2018 Dec;46(14):3471-3479. doi: 10.1177/0363546518807908. Epub 2018 Nov 12. PMID 30419178
- [Background] Carkci E, Polat AE, Gurpinar T. The frequency of reduction loss after arthroscopic fixation of acute acromioclavicular dislocations using a double-button device, and its effect on clinical and radiological results. J Orthop Surg Res. 2020 Apr 8;15(1):136. doi: 10.1186/s13018-020-01674-x. PMID 32268914
- [Background] Ladermann A, Denard PJ, Collin P, Cau JBC, Van Rooij F, Piotton S. Early and delayed acromioclavicular joint reconstruction provide equivalent outcomes. J Shoulder Elbow Surg. 2021 Mar;30(3):635-640. doi: 10.1016/j.jse.2020.06.026. Epub 2020 Jul 7. PMID 32650071